CLINICAL TRIAL: NCT03180437
Title: Safety and Efficiency of IRE Plus γδ T Cell Against Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Jinan University Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gd T cell and Pancreatic Ca
Record Dates: First submitted 2017-05-19; First posted 2017-06-08 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-07

CONDITIONS: Pancreatic Cancer
Keywords: Immunotherapy; γδ T Cell; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): In this group, the patients will receive IRE surgery to control the local tumor under CT .
  Interventions: Procedure: IRE surgery
- Group B (Experimental): In this group, the patients will receive multiple high-activity γδ T cell immunotherapies and IRE surgery
  Interventions: Biological: IRE plus γδ T cells

INTERVENTIONS:
Procedure: IRE surgery — IRE surgery will be used in local tumor
  Arms: Group A
Biological: IRE plus γδ T cells — Combination IRE surgery and γδ T cell will be used in Pancreatic Cancer
  Arms: Group B

SUMMARY:
In this study, effects of γδT cells on human Pancreatic Cancer in combination with tumor reducing surgery, for example IRE going to be investigated.

DETAILED DESCRIPTION:
Pancreatic tumor will be removed using tumor reducing surgery such as IRE. PBMC of the healthy donor will be separated from peripheral blood. After making them potential cancer killer γδ T Cell, they will be infused to the patients as an immunotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. age: >18 years
2. participants older than 18 years with either LAPC according to the American Joint Committee on Cancer (AJCC) criteria or isolated local recurrence with a maximum tumor diameter of 5 cm were considered eligible after pathologic confirmation
3. will receive IRE, gd Tcells
4. life expectancy: more than 3 months
5. ability to understand the study protocol and a willingness to sign a written informed consent document
6. adequate liver and renal function were required
7. intolerant or refused to chemotherapy or to chemotherapy

Exclusion Criteria:

1. patients with other kinds of cancer
2. history of coagulation disorders or anemia
3. heart disease and diabetes
4. history of epilepsy, severe coronary disease, a history of level 3 hypertension，myelosuppression, autoimmune disease
5. a performance status score of >2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
PFS | 2 years
  PFS was defined as the interval between treatment initiation and local relapse
OS | 2 year
  OS was calculated as the interval from treatment initiation to death.

SECONDARY OUTCOMES:
Tumor size | 3 months
  The tumor responses of the enrolled patients were assessed by CT in accordance with RECIST v1.1.Institute Common Terminology Criteria for Adverse Events (v4.0).
CTC | 3 months
  The absolute number of CD45-CK+ CD326+ cells was used to quantitate the CTC levels.
CA 19-9 | 3 months
  The serum concentrations of CA19-9 were evaluated by a chemiluminescent immunoassay before treatment and 90 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jibing Chen, PhD, Principal Investigator — Biological treatment center in Fuda cancer hospital Guangzhou
Locations (1):
- Biotherapy center in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lin M, Zhang X, Liang S, Luo H, Alnaggar M, Liu A, Yin Z, Chen J, Niu L, Jiang Y. Irreversible electroporation plus allogenic Vgamma9Vdelta2 T cells enhances antitumor effect for locally advanced pancreatic cancer patients. Signal Transduct Target Ther. 2020 Oct 23;5(1):215. doi: 10.1038/s41392-020-00260-1. PMID 33093457